CLINICAL TRIAL: NCT05365750
Title: COVID-19 Antibody and Reinfection Study
Status: Completed | Type: Observational
Sponsor: Kaiser Permanente (Other)
Responsible Party: Principal Investigator, Ingrid Binswanger, Senior Investigator, Kaiser Permanente
Other Study IDs: 1589316-19
Record Dates: First submitted 2022-05-05; First posted 2022-05-09 (Actual); Results first posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-08

CONDITIONS: COVID-19 Testing
Keywords: SARS-CoV-2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case: Case patients were drawn from a random sample of individuals who were enrolled in KPCO's health plan had suspected or confirmed SARS-CoV-2 infection and a random stratified sample of the general KPCO membership with similar age, gender, race/ethnicity and co-morbidities as case group. Within the cohort, case patients had a SARS-CoV-reinfection, defined as a positive SARS-CoV-2 RNA test ≥ 90 days after the first positive RNA test.
- Control: Control patients were drawn from a random sample of individuals who were enrolled in KPCO's health plan had suspected or confirmed SARS-CoV-2 infection and a random stratified sample of the general KPCO membership with similar age, gender, race/ethnicity and co-morbidities as case group. Within the cohort, control patients had no evidence of a SARS-CoV-reinfection during the period of interest.

SUMMARY:
The goal of this study is to establish a cohort of Kaiser Permanente Colorado (KPCO) members who have and have not had COVID-19 infection for serial antibody testing and PCR testing to:

1. Quantify antibody titers among participants over 9 months.
2. Determine the rates of asymptomatic, mild, and severe recurrent infection among participants with prior COVID-19.
3. Examine association between antibody titer levels and risk of recurrent infection using a case control analysis nested in the cohort.

DETAILED DESCRIPTION:
In this study, the Kaiser Permanente Colorado (KPCO) Institute for Health Research (IHR) will evaluate SARS-CoV-2 IgG antibody titers over time among individuals with evidence of prior infection, and correlate antibody titers with risk of recurrent infection. The investigators will identify KPCO members who have and have not had prior infection, enroll them into a cohort study, conduct serial surveys for new COVID-19 symptoms, and facilitate serial viral and antibody testing.

All laboratory testing procedures and clinical management of participants will be conducted by KPCO operations. The research team will identify participants, obtain consent, administer surveys to assess COVID-19 symptoms, and direct patients to the appropriate testing. Health outcomes on cohort participants will be tracked with survey data on symptoms, clinical and utilization data from the KPCO electronic health record (e.g., hospitalization), and laboratory data (e.g., viral test results).

This research-operations partnership strategy will generate data to better understand the implications of positive antibody titers to this novel pathogen.

ELIGIBILITY:
Inclusion criteria are Kaiser Permanente Colorado health plan members, with a valid email address or phone number in the electronic health record and not on the Do Not Call List for research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study cohort will include individuals who are enrolled in Kaiser Permanente Colorado's health plan. Individuals will be selected who have evidence of prior SARS CoV-2 infection and random samples of the general KPCO membership of similar demographic characteristics who appear not to have had SARS CoV-2 infection.
Sampling Method: Probability Sample
Enrollment: 4235 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2024-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ingrid Binswanger, MD, MPH, MS, Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Permanente, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Binswanger IA, Narwaney KJ, Barrow JC, Albers KB, Bechtel L, Steiner CA, Ann Shoup J, Glanz JM. Association between severe acute respiratory syndrome coronavirus 2 antibody status and reinfection: A case-control study nested in a Colorado-based prospective cohort study. Prev Med Rep. 2023 Dec 1;37:102530. doi: 10.1016/j.pmedr.2023.102530. eCollection 2024 Jan. PMID 38205171
- See also: Publication — https://doi.org/10.1016/j.pmedr.2023.102530

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited into a cohort from the health plan membership from June 2020 to March 2021 using text message and emails linked to online consent documents. From this cohort, we conducted a nested case control analysis in which participants with the outcome were compared to participants without the outcome.
Pre-assignment Details: As is standard in a nested case-control study, the cohort is used to identify a sufficient sample to conduct the case-control analysis, in which people with the outcome of interest are compared with people who did not have the outcome. The protocol section describes the recruited cohort (n=4235) and the results section describe participants in the case-control (n=1114). Participants not in the case-control (n=3121) are not in the participant flow because their data were not analyzed.
Groups:
- Case Patients Nested Within the Cohort: Case patients had a reinfection, defined as a positive SARS-CoV-2 RNA test ≥ 90 days after the first positive RNA. Case patients had serology completed between the infections.
- Control Patients Nested Within the Cohort: Control patients had a primary infection and serologic tests that were conducted between the primary infection and the index date. A control patient could be matched to more than one case patient if they had more than one eligible serologic test. Case patients were 1:20 matched to controls.
Period: Overall Study
Arm/Group | Case Patients Nested Within the Cohort | Control Patients Nested Within the Cohort
Started | 80 | 1034
Completed | 80 | 1034
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The analysis population is cases (n=80) and controls (n=1034) within a cohort (n=4235).
Groups:
- Total: Total of all reporting groups
Arm/Group | Case Patients Nested Within the Cohort | Control Patients Nested Within the Cohort | Total
Number analyzed (Participants) | 80 | 1034 | 1114
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.7 (12.7) | 54.4 (11.9) | 54.3 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 761 | 821
  Male | 20 | 273 | 293
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 32 | 252 | 284
  Not Hispanic or Latino | 48 | 782 | 830
  Unknown or Not Reported | 0 | 0 | 0
Negative serologic test [Number; unit: participants] | 12 | 77 | 89

OUTCOME MEASURES:

1. Primary Outcome: Reinfection With SARS-CoV-2
Description: In this case-control analysis, case patients were participants with the outcome of reinfection. The date of reinfection was the index date. Control patients were those with a primary infection but without the outcome reinfection by the index date. The case and control participants were compared with respect to a seronegative test result (exposure) after primary infection and closest in time to the index date. Because the cases and controls were selected on the basis of the outcome, the seronegative result is listed below by case and control status.
Time Frame: Through the completion of the study analytic period, an average of 6 months
Population: Study cohort members with a primary SARS-CoV-2 infection
Measure: Count of Participants; unit: Participants
Groups:
- Case Patients: Participants with reinfection, defined as a positive SARS-CoV-2 RNA test ≥ 90 days after the first positive RNA test
- Control Patients: Participants without reinfection
Arm/Group | Case Patients | Control Patients
Number analyzed (Participants) | 80 | 1034
Participants
  Seronegative test results | 12 | 77
  Seropositive test results | 68 | 957

ADVERSE EVENTS:
Time Frame: Through the completion of the study analytic period, an average of 6 months
Description: This was not a clinical trial but a nested case-control study. Following IRB approved procedures, we collected adverse events (AEs) and serious adverse events (SAE) related to study procedures (surveys, testing), related and un-related COVID-related hospitalizations (SAEs), and related and unrelated all-cause deaths (SAEs). Other unrelated AEs and SAEs were not collected as part of this study focused on COVID. AEs and SAEs and deaths are reported for case-control participants.
Arm/Group | Case Patients Nested Within the Cohort | Control Patients Nested Within the Cohort
All-Cause Mortality (participants affected / at risk) | 0/80 | 0/1034
Serious Adverse Events (participants affected / at risk) | 0/80 | 0/1034
Other Adverse Events (participants affected / at risk) | 0/80 | 0/1034

LIMITATIONS AND CAVEATS:
Adherence to the study's testing guidance was inconsistent. We encouraged regular on-site testing but may not have captured some home-based testing results. Variable sensitivity and specificity of different serologic tests could have influenced our results. Variable sero-reversion rates across tests could have been due to variable lengths of time between the primary infection and testing. The definition of a reinfection used could have identified viral persistence.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-01): https://cdn.clinicaltrials.gov/large-docs/50/NCT05365750/Prot_SAP_000.pdf